CLINICAL TRIAL: NCT04846322
Title: Pathway to Detection & Differentiation of Delirium & Dementia in the Emergency Department
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000029490; U54AG063546 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-04-15 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Impairment; Emergency Care; Dementia; Delirium
Keywords: delirium
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ED delirium & dementia screening & outpatient referral: Routine ED screening for delirium and memory problems with referral for outpatient assessment of cognitive impairment.
  Interventions: Diagnostic Test: PD4ED 3-step intervention (ED assessment, outpatient assessment, Brain health plan)

INTERVENTIONS:
Diagnostic Test: PD4ED 3-step intervention (ED assessment, outpatient assessment, Brain health plan) — 1. ED assessment for suspected dementia.
  2. positive ED patients referred for outpatient clinic cognitive impairment assessment.
  3. positive clinic patients referred to primary care with brain health patient plan.

SUMMARY:
This is an observational study of the pragmatic implementation of an ED screening, outpatient referral, and care coordination process for older ED patients who may have UCID.

DETAILED DESCRIPTION:
Embedded pragmatic, implementation pilot that incorporates training, ED assessment for delirium and dementia risk, referral of ED patients with undiagnosed cognitive impairment and dementia for primary care feedback and care recommendations. This pilot would gather observational data evaluating the feasibility of incorporating cognitive impairment screens into routine ED delirium assessments, and developing optimal work flow for identifying and referring ED patients with suspected (undiagnosed) dementia for confirmatory evaluation and care coordination.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 65 or older
* Discharged from the adult ED at YNHH or the ED at NMH

Exclusion Criteria:

* Documented or known history of dementia
* Alcohol/substance intoxication while in the ED
* Non-English or Non-Spanish speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All community dwelling ED patients 65 years of age or older seen in the Yale New Haven Health System (YNHHS) St. Raphael's Campus (SRC) ED or Northwestern Memorial Hospital (NMH) ED.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ula Hwang, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Northwestern, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- ED Delirium & Dementia Screening & Outpatient Referral: Routine ED screening for delirium and memory problems with referral for outpatient assessment of cognitive impairment.
  PD4ED 3-step intervention (ED assessment, outpatient assessment, Brain health plan): 1. ED assessment for suspected dementia.
  2. positive ED patients referred for outpatient clinic cognitive impairment assessment.
  3. positive clinic patients referred to primary care with brain health patient plan.
Period: Overall Study
Arm/Group | ED Delirium & Dementia Screening & Outpatient Referral
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ED Delirium & Dementia Screening & Outpatient Referral
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 82 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 29
  White | 60
  Asian | 5
  Other | 1
  Unknown or not reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 100
ED delirium diagnosis [Count of Participants; unit: Participants] | 9
ED Confusion Assessment Method (CAM) Positive [Count of Participants; unit: Participants] — CAM is a standardized evidence-based tool that enables non-psychiatrically trained clinicians to identify and recognize delirium quickly and accurately in both clinical and research settings. A positive score is based on the presence of two major criteria and at least one of the minor criteria.
  Participants | 7
Chronic Conditions [Count of Participants; unit: Participants]
  High blood pressure | 73
  Stroke | 14
  TBI | 2
  PVD | 4
  Renal failure | 14
  Diabetes | 33
Emergency Severity Index Level [Mean (Standard Deviation); unit: score on a scale] — Severity of the emergency triage score while in ED, 1 = acute to 5 = non-urgent
  score on a scale | 2.7 (0.7)
Emergency Department (ED) memory screen [Count of Participants; unit: Participants] — Percent of participants that had a memory screen while in the ED
  Participants | 41
Dementia or Alzheimer's self report [Count of Participants; unit: Participants] — Dementia or Alzheimer's listed by participant per problem list at the time of ED visit
  Participants | 20
Top 3 chief complaints per participants self report [Count of Participants; unit: Participants] — Top 3 chief complaints per participants self report at time of ED visit
  Participants
    Altered mental status | 21
    Fall | 17
    Abdominal pain | 7
ED Disposition [Count of Participants; unit: Participants]
  Discharged | 88
  Admitted | 4
  Observation | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Confirmed Delirium or Dementia
Description: percentage of patients discharged from ED positive for delirium or dementia among total number of patients 65+
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | ED Delirium & Dementia Screening & Outpatient Referral
Number analyzed (Participants) | 88
percentage of participants | 30.8

2. Primary Outcome: Rates of Outpatient Assessment Referral of Patients With Suspected Dementia
Description: number of patients with appointment to Alzheimer's Dementia Centers or geriatrics outpatient clinic / number of patients given information sheet or referred to outpatient clinic
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ED Delirium & Dementia Screening & Outpatient Referral
Number analyzed (Participants) | 100
Participants | 26

3. Primary Outcome: Number of Participants Diagnosed With Dementia Among Those With Completed Outpatient Assessment
Description: number of patients diagnosed with dementia (all categories) among those that completed the outpatient assessment
Time Frame: Up to 100 days from ED discharge
Population: 19 completed the outpatient assessment
Measure: Count of Participants; unit: Participants
Arm/Group | ED Delirium & Dementia Screening & Outpatient Referral
Number analyzed (Participants) | 19
Participants | 15

4. Primary Outcome: Rates of Connection With Primary Care
Description: number of patients with PCP follow-up about brain health plan of the number of patients with outpatient confirmation of Dementia or MCI
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | ED Delirium & Dementia Screening & Outpatient Referral
Number analyzed (Participants) | 100
Participants | 19

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) evaluated retrospectively via chart review during 90-day of follow-up period.
Arm/Group | ED Delirium & Dementia Screening & Outpatient Referral
All-Cause Mortality (participants affected / at risk) | 2/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 6/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ED Delirium & Dementia Screening & Outpatient Referral (N=100)
Mood alteration (Psychiatric disorders) | 3 — Depression
Mood alteration (Psychiatric disorders) | 3 — Anxiety

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT04846322/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04846322/ICF_001.pdf